CLINICAL TRIAL: NCT06939244
Title: Investigating the Effects of Krill Oil on the Recovery From Muscle Damaging Exercise: a Randomised Controlled Trial
Acronym: KORE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Stuart Gray, Professor Stuart Gray, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KORE
Record Dates: First submitted 2025-03-25; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-03

CONDITIONS: Looking at the Effects of Krill Oil Supplementation on Recovery From Muscle-damaging Exercise
Keywords: Omega-3; Exercise; Muscle
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Krill oil Supplement (Experimental): 2g of Krill oil per day
  Interventions: Dietary Supplement: Krill oil
- Mixed Vegetable Oil (Placebo Comparator): 2g of Mixed Vegetable Oil per day
  Interventions: Dietary Supplement: Krill oil

INTERVENTIONS:
Dietary Supplement: Krill oil — Krill oil supplement

SUMMARY:
1. What will happen to me if I take part?

All study visits will be at the University of Glasgow main campus within the Sir James Black building.

Initial visit (duration 1 hours)

We will ask that for each study visit you come to the laboratory with clothing suitable to exercise in (loose shorts) for your own comfort and to also make it easier for us to complete certain measurements where access to upper legs will be necessary. Changing facilitates will be provided on-site. After the screening process, your physical activity and your diet will be assessed via questionnaires. We will then familiarise you with the physical function tests and neuromuscular measurements.

Visit 2 (duration 1 hours)

Before the remaining study visits in the morning, you will be asked to arrive at the laboratory after an overnight fast (no food or caffeinated/calorific beverages from 10pm), and without having done intense exercise for two days prior to the visit. Upon arriving in the laboratory, we will collect a blood sample (after which we will provide you with a snack), and measure your body composition, muscle size, muscle strength and physical function. You will then be familiarised with the resistance training protocol, and we will determine your maximum strength for two leg exercises. After these measurements are completed, we will randomly assign you to consumed 2g/day of either krill oil or a mixed vegetable oil.

Visit 3 (duration 3 hours)

After 8 weeks of supplementation, you will attend for a third study visit. This will involve a blood sample and repeating the same measures from the baseline visit with the addition of a measurement of soreness in the upper legs. We will then ask you to complete muscle-damaging exercises consisting of a warm-up of 5 minutes of downhill walking (5% decline at a self selected speed between 3-6 km/h) followed by 4 sets of machine exercises of both leg kicking and leg pushes. These leg exercises will be performed at ~70% of your maximum strength and we will ask you to perform as many repetitions as you can, with the last two sets of each exercise also consisting of 4 extra lowering repetitions. Five minutes and 60 minutes following the muscle-damaging exercise, all the measurements, including blood samples, will be repeated.

Visit 4 (duration 1 hours)

Two days after visit 3, we will once again repeat the measures taken on visit 3 for a final time.

Measurements

Blood sample: A blood sample (15ml) will be collected from a vein in your arm by a trained member of the research team.

Muscle size: We will use an ultrasound to assess muscle thickness of one of the muscles on the outside of your legs.

Muscle strength: You will sit in a chair with your legs at a 90-degree angle. A strap will be placed around the right ankle which will be connected to a force sensor and three sticky surface electrodes will be placed on your thigh. We will then ask you to contract as hard as you can with the leg fixed in position, and we will record the force for 5 seconds. You will perform 3 contractions, with a 1min rest between contractions. After the maximal contractions, will be ask you to contract at 20, 35 and 50% of your maximal effort for 15 seconds so that we can record electrical activity in your muscle. We will then stimulate a contraction with a small electrical current at rest and during a maximal contraction.

We will also measure grip strength, making 3 measures from each hand. We will measure your strength on exercise machines, for both leg kicking and leg pushing. Following a warm-up, the weights on each machine will be progressively increased in until you cannot do any more.

Physical function: We will ask you to rise from a chair 5 times and to walk a distance of 4 metres and record how long this takes. We will also ask you to stand for 10 seconds with your legs in 3 different positions. These will be demonstrated to you before you do this.

Body composition: We will measure total fat and lean mass using bioelectrical impedance analysis.

Soreness: We will ask you to mark on a line how sore your muscle feels to measure muscle soreness before and immediately after the muscle damage protocol in two different tests. In the first test, we will apply a fixed, moderate amount of pressure on your thigh and we will ask you how sore it feels; in the second test, we will apply an increasing amount of pressure until on your thigh until you tell us it feels sore.

ELIGIBILITY:
Inclusion Criteria:

* Be 60 years old or older
* Have a BMI of less than 30kg/m2
* Participating in resistance-type exercise for less than 1h per week

Exclusion Criteria:

* Diabetes
* Severe cardiovascular disease defined as arrythmia, valve disease, coronary artery disease, heart failure, peripheral arterial disease, cerebrovascular disease, congenital heart disease or myocardial infarct.
* Seizure disorders
* Uncontrolled hypertension (blood pressure higher than 150/90mmHg at baseline measurement)
* Cancer or cancer that has been in remission for less than 5 years
* Ambulatory impairments limiting the ability to perform muscle function assessments
* Dementia
* Taking medications known to affect muscle (like steroids)
* Having an implanted electronic device (such as a pacemaker, defibrillator, or insulin pump)
* Allergies to seafood
* Regular consumption of more than one portion of oily fish per week

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Muscle soreness (Habitual Soreness) | 0 to 48 hours (Post Intervention)
  Visual Analogue Scales will be used to measure muscle soreness before and immediately after the muscle damage protocol. This assessment with a visual analogue scale will be done after asking the participant to sit down and stand up from a chair twice to determine muscle soreness during habitual physical activity.
Muscle soreness (Pain Pressure Threshold) | 0 to 48 hours (Post Intervention)
  Visual Analogue Scales will be used to measure muscle soreness before and immediately after the muscle damage protocol. This assessment, with a visual analogue scale and handheld soreness pressure algometer, will determine the pressure threshold required to cause soreness and will be taken at the site which is 10% of the circumference laterally from the mid-point between the iliac crest and the top of the patella.
Muscle soreness (5kg/cm2) | 0 to 48 hours (Post Intervention)
  Visual Analogue Scales will be used to measure muscle soreness before and immediately after the muscle damage protocol. This assessment with a visual analogue scale and handheld soreness pressure algometer will be in response to 5kg/cm2 of pressure delivered at 10% of the circumference laterally from the mid-point between the iliac crest and the top of the patella.

SECONDARY OUTCOMES:
Fatty Acid Composition | From enrollment to the end of treatment at 8 weeks
  A venous blood sample (15ml) will be collected by a trained member of the research team from an antecubital vein and analysed for erythrocyte fatty acid profile.
Muscle size | From enrollment to the end of treatment at 8 weeks
  We will use ultrasound to assess muscle thickness of the vastus lateralis muscle using B-mode ultrasound with the participants in a supine position. This will also be an indirect measure of muscle damage from cell swelling. The site of the measurement will be 10% of the circumference laterally from the mid-point between the iliac crest and the top of the patella.
Knee Extensor Strength | From enrollment to the end of treatment at 8 weeks
  We will measure muscle strength of the knee extensor muscles during a maximal voluntary contraction (MVC) at a 90-degree angle
Fat mass | From enrollment to the end of treatment at 8 weeks
  Fat mass will be determined by bioelectrical impedance analysis.
Grip Strength | From enrollment to the end of treatment at 8 weeks
  Grip strength will be determined pre- and post the 8-week supplementation period and will be measured with a hand grip dynamometer.
Gait Speed | From enrollment to the end of treatment at 8 weeks
  Gait speed will be assessed as a measurement of physical function.
Balance | From enrollment to the end of treatment at 8 weeks
  Balance will be assessed by the duration at which they can balance with three separate foot positions
Chair rise time | From enrollment to the end of treatment at 8 weeks
  Chair rise time will be assessed by the time it takes for the participant to sit down and sit down 5 times
Lean Mass | From enrollment to the end of treatment at 8 weeks
  Lean mass will be determined by bioelectrical impedance analysis.
Muscle Fiber Conduction Velocity | From enrollment to the end of treatment at 8 weeks
  Muscle Fiber Conduction Velocity will be assessed by HD-EMG at three different intensities of MVC. 20%, 35% and 50%.
Voluntary Activation | From enrollment to the end of treatment at 8 weeks
  Voluntary Activation (VA) is assessed using neuromuscular measurements during muscle strength testing, involving both measurement of force and electrical stimulation of the femoral nerve
Creatine Kinase | 0 to 48 hours (Post Intervention)
  Creatine Kinase will be assessed by a blood draw prior to, immediately following, 1 hour after and 48 hours after resistance exercise
Muscle Size | 0 to 48 hours (Post Intervention)
  We will use ultrasound to assess muscle thickness of the vastus lateralis muscle using B-mode ultrasound with the participants in a supine position. This will also be an indirect measure of muscle damage from cell swelling. The site of the measurement will be 10% of the circumference laterally from the mid-point between the iliac crest and the top of the patella.
Knee Extensor Strength | 0 to 48 hours (Post Intervention)
  We will measure muscle strength of the knee extensor muscles during a maximal voluntary contraction (MVC) at a 90-degree angle
Gait Speed | 0 to 48 hours (Post Intervention)
  Gait speed will be assessed as a measurement of physical function.
Balance | 0 to 48 hours (Post Intervention)
  Balance will be assessed by the duration at which they can balance with three separate foot positions
Chair rise time | 0 to 48 hours (Post Intervention)
  Chair rise time will be assessed by the time it takes for the participant to sit down and sit down 5 times
Muscle Fiber Conduction Velocity | 0 to 48 hours (Post Intervention)
  Muscle Fiber Conduction Velocity will be assessed by HD-EMG at three different intensities of MVC. 20%, 35% and 50%.
Voluntary Activation | 0 to 48 hours (Post Intervention)
  Voluntary Activation (VA) is assessed using neuromuscular measurements during muscle strength testing, involving both measurement of force and electrical stimulation of the femoral nerve

CONTACTS AND LOCATIONS:
Locations (1):
- University of Glasgow, Glasgow, Other, United Kingdom

IPD SHARING:
Plan to Share IPD: No